CLINICAL TRIAL: NCT06888466
Title: Personalised HeartCare: Poligenic Risk Scores Disclosure for Cardiovascular Prevention and Behavioral Change
Brief Title: Personalised HeartCare: Poligenic Risk Scores Disclosure for Cardiovascular Prevention
Acronym: PHC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Stefania Boccia, Full Professor of Hygiene and Preventive Medicine, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6732
Record Dates: First submitted 2025-02-24; First posted 2025-03-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular prevention; Polygenic Risk Score
MeSH Terms: conditions — Cardiovascular Diseases; Genetic Risk Score

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRS (Experimental): Lifestyle coaching and genetic intervention: calculation of the Polygenic Risk Score (PRS)
  Interventions: Behavioral: The result of the Polygenic Risk Score will be communicated to the patient with the aim of encouraging a change in behavior

INTERVENTIONS:
Behavioral: The result of the Polygenic Risk Score will be communicated to the patient with the aim of encouraging a change in behavior — Blood samples collected for the calculation of the genetic predisposition profile for Cardiovascular risk will be used for DNA extraction and genotyping, and the PRS will subsequently be calculated. Based on the results, individuals will be classified into three main CVD risk categories (high risk, intermediate risk, low risk)

SUMMARY:
The goal of this clinical trial is to evaluate whether the disclosure of Polygenic Risk Scores (PRS) combined with personalized coaching on risk factors can lead to significant improvements in lifestyle behaviors among staff members at Fondazione Policlinico Universitario Agostino Gemelli IRCCS. The study includes staff members from Fondazione Policlinico Universitario Agostino Gemelli IRCCS, enrolled at the outpatient clinics of the Cardiology Department.

Main Research Questions:

1. Does receiving PRS disclosure and personalized coaching lead to significant improvements in lifestyle behaviors compared to baseline measurements?
2. How do different levels of genetic predisposition to cardiovascular diseases (CVD) impact behavioral changes following intervention? This is a single arm, pre-post clinical trial.

Participant will:

* Undergo genetic testing to assess their Polygenic Risk Score for CVDs
* receive personalized, in-person consultation with a medical cardiologis, together with and individualized recommendations for CVD prevention based on PRS results and traditional risk factors.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy of disclosing cardiovascular genetic risk-specifically through the Polygenic Risk Score (PRS)-in promoting the adoption of healthier lifestyle behaviors.

The enrollment period will last 18 months, with each participant taking part in the study for six months. There are three key time points in the study, T0 or baseline (enrollment phase), T1 or disclosure visit, T2 or final visit at six months. At enrollment, participants will be classified into risk categories based on cardiovascular risk using the SCORE-2 or SCORE 2-OP tool. Individuals with a SCORE-2 <10% or SCORE 2-OP <15% will be invited to join the PHC pilot study.

Study Procedures Baseline Evaluations (T0)

After providing informed consent specific to the PHC study, participants will undergo the following assessments:

* Personal and Family History, Socioeconomic and Professional Status, and Demographic Information: a structured questionnaire will be administered at T0 to collect data on medical history, family history, socioeconomic and professional status, and demographic information.
* LE'8 Lifestyle Questionnaire: the Life's Essential 8 (LE'8) lifestyle questionnaire will be administered at T0 and T2. It generates a lifestyle score that categorizes participants into three groups: favorable, intermediate, or unfavorable. Validated in European populations and widely used in clinical studies, the scale ranges from 0 to 100.
* Medical Examination: includes biometric measurements such as BMI, body circumference, heart rate, and blood pressure.
* Blood Test Results: participants will provide recent blood test results (within the last six months) for lipid profiles, C-reactive protein (CRP), and glucose or hemoglobin A1c, which will be used to calculate the SCORE-2/SCORE 2-OP score.
* Blood Sampling: blood samples will be collected to perform genetic testing and assess cardiovascular disease risk through Polygenic Risk Scores (PRS).
* Anxiety Assessment (GAD-7): Participants will complete the Generalized Anxiety Disorder (GAD-7) questionnaire at T0 and T2 to assess anxiety levels.
* Work Ability: Participants will complete the Work Ability Index (WAI) questionnaire at T0 and T2 to assess their work ability.

Disclosure Visit (T1)

Approximately one month after T0, participants will undergo a telematic follow-up visit, during which:

* Their lifestyle score will be explained.
* Personalized preventive advice will be provided to encourage healthier lifestyle changes.
* PRS results will be disclosed, along with the corresponding genetic risk category (high, intermediate, or normal).

Follow-up Visit (T2)

Six months after the disclosure visit (T1), participants will undergo a comprehensive follow-up evaluation, which will include:

* Lifestyle Questionnaire: Assessment of lifestyle changes since T0.
* Recalculation of Lifestyle Category: Based on updated responses to the lifestyle questionnaire.
* Biometric Measurements: Includes weight, BMI, body circumference, heart rate, and blood pressure.
* Acceptability Questionnaire: Both participants and medical professionals will complete a questionnaire on the acceptability of the intervention.
* Preferences on Technology Use: A questionnaire assessing participants' values and preferences regarding new technologies in healthcare.
* Genetic Testing Reaction (FACToR): A modified version of the MICRA questionnaire will be used to evaluate participants' reactions to genetic testing.
* WAI questionnaire to evaluate their work ability

ELIGIBILITY:
Inclusion criteria

* Traditional cardiovascular risk: The risk will be assessed using SCORE 2 (low risk < 2.5%, moderate risk between 2.5% and 5%, high risk between 5% and 10%) or SCORE 2-OP (moderate risk < 7.5%, high risk between 7.5% and 15%).
* Blood tests: Participants must have had blood tests performed within the past 6 months.
* Age: Participants must be at least 40 years old.

Exclusion Criteria

* Very high cardiovascular risk, as measured by SCORE 2 (very high risk > 10%) or SCORE 2-OP (very high risk > 15%).
* Diabetes.
* Familial hypercholesterolemia.
* Previous cardiovascular events or established CVD

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in the lifestyle profile | From enrollment to the final follow-up at 6 months.
  The lifestyle category will be measured using the Life's Essential 8 tool. A change will be considered achieved if there is a shift towards a more favorable lifestyle category at final follow-up at 6 months compared to baseline. The overall score ranges from 0 to 100, and the categories are three:
  * 0-49:Poor cardiovascular health
  * 50-79: Intermediate cardiovascular health
  * 80-100: Optimal cardiovascular health

SECONDARY OUTCOMES:
Change in the LDL-Cholesterol | From enrollmentto the final follow-up at 6 months
  LDL-cholesterol (LDL-C) will be measured in mg/dL from fasting blood samples. The outcome will be defined as the change in LDL-C levels between baseline (enrollment) and final follow-up at 6 months.
Change in cardiovascular disease risk | From enrollment to the final follow-up at 6 months.
  The CVD risk of participants will be estimated using the SCORE2 (for individuals aged 40-69 years) and SCORE2-OP (for individuals aged ≥70 years) charts. A change will be defined as a shift towards a lower estimated risk at 6-month follow-up compared to baseline. The SCORE2 and SCORE2-OP classify individuals into four categories of 10-year risk of CVD events:
  * Low to moderate risk: <5% (SCORE2, age 40-49), <7.5% (age 50-69), <10% (SCORE2-OP, age ≥70)
  * High risk: 5-10% (age 40-49), 7.5-15% (age 50-69), 10-20% (age ≥70)
  * Very high risk: >10% (age 40-49), >15% (age 50-69), >20% (age ≥70)
Smoking habit modification | From enrollment to the final follow-up at 6 months.
  Number of participants who have quit or reduced smoking at the final follow-up at 6 months compared to baseline.
Change in Alcohol Consumption | From enrollment to the final follow-up at 6 months.
  Number of participants who have quit or reduced alcohol consumption at the final follow-up at 6 months compared to baseline.
Anxiety | Measured at enrollment and again one month after receiving PRS results.
  Level of anxiety before and after the administration of Polygenic Risk Score testing and the disclosure of results, measured through the GAD-7 questionnaire. The total score ranges from 0 to 21, with higher scores indicating greater anxiety severity (0-4: Minimal anxiety; 5-9: Mild anxiety; 10-14: Moderate anxiety; 15-21: Severe anxiety)
Reaction to genetic test | Measured 1 month after the baseline visit
  Evaluation of the psychosocial impact of returning genomic findings to patients, through the FACToR questionnaire. It consists of 12 items divided into four subscales: negative emotions, positive emotions, uncertainty, and privacy concerns.
Change in dietary habits score (Life's Essential 8 questionnaire) | From enrollment to the final follow-up at 6 months
  Dietary habits will be assessed using the diet component of the Life's Essential 8 questionnaire. Scores range from 0 (poor) to 100 (ideal), based on frequency and quality of food intake (e.g., fruit/vegetable consumption, whole grains, sugar-sweetened beverages, fish, sodium intake). A higher score indicates healthier dietary habits. The outcome will be defined as the change in diet score from baseline to 6-month follow-up.
Change in physical activity score (Life's Essential 8 questionnaire) | From enrollment to the final follow-up at 6 months
  Physical activity will be assessed using the activity component of the Life's Essential 8 questionnaire. Scores range from 0 (poor) to 100 (ideal), based on self-reported weekly minutes of moderate-to-vigorous physical activity. A higher score indicates more favorable physical activity behavior. The outcome will be defined as the change in activity score from baseline to 6-month follow-up.
Accetability of PRS testing | Measured at 6 months at the final follow-up
  Acceptability of PRS testing will be assessed with a 7-item structured questionnaire completed by clinicians. Each item is rated on a 1-4 Likert scale (1 = strongly disagree, 4 = strongly agree). The outcome will be defined as the proportion of clinicians and of patients reporting high acceptability (scores of 3-4).
Feasibility of the PRS testing | Measured at 6 months at the final follow-up
  Feasibility of integrating PRS testing into the clinical care pathway will be evaluated using an 11-item questionnaire administered to physicians. Responses are rated on a 1-4 Likert scale (1 = strongly disagree, 4 = strongly agree). The endpoint will be the proportion of clinicians reporting high acceptability (scores of 3-4) of PRS testing.
Change in self-assessed work ability (Work Ability Index, WAI) | From enrollment to the final follow-up at 6 months.
  Work ability will be evaluated among employed participants using the Work Ability Index (WAI). The questionnaire consists of approximately 60 items across seven subscales: (1) current work ability compared with lifetime best, (2) work ability in relation to job demands, (3) number of current diseases diagnosed by a physician, (4) estimated work impairment due to diseases, (5) sick leave during the past year, (6) own prognosis of work ability in two years, and (7) mental resources.
  The outcome will be defined as the change in WAI total score from baseline to 6-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento Universitario di Scienze della Vita e Sanità Pubblica, Roma, Italia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: EU Health Policy — https://health.ec.europa.eu/eu-health-policy/overview_en
- See also: PNRR - Governo Italiano Presidenza del Consiglio dei Ministri — https://www.governo.it/it
- See also: Next Generation Italia, approvato il piano del Governo - Next Generation Italia, approvato il piano del Governo — https://innovazione.gov.it
- See also: Personalised Medicine - European Commision — https://european-union.europa.eu/index_it